CLINICAL TRIAL: NCT02838030
Title: Efficacy of the Combination of Acetylsalicylic Acid and L-arginine to Prevent Preeclampsia in Pregnant High Risk
Brief Title: Efficacy of Aspirin and L-arginine in High Risk Preeclamptic
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University of Guadalajara (Other)
Collaborators: PhD Ernesto Javier Ramírez Lizardo (Unknown); PhD Sylvia Elena Totsuka Sutto (Unknown); PhD Fernando Grover Páez (Unknown); MD Diego Hernández Molina (Unknown)
Responsible Party: Principal Investigator, Leonel Garcia Benavides, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ECAALA
Record Dates: First submitted 2016-05-26; First posted 2016-07-20 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: High Risk Pregnancy
Keywords: Preeclampsia; L-arginine
MeSH Terms: conditions — Pre-Eclampsia | interventions — Arginine; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acetylsalicylic acid and L-arginine (Experimental): acetylsalicylic acid 75 mg every 24 hours from the 12th week of pregnancy and L-arginine 3 gr every 8 hours from the 20th week of pregnancy to pregnancy termination
  Interventions: Drug: L-arginine; Drug: acetylsalicylic acid
- acetylsalicylic acid and placebo (Placebo Comparator): acetylsalicylic acid 75 mg every 24 hours from the 12th week of pregnancy and placebo 3 gr every 8 hours from the 20th week of pregnancy to pregnancy termination
  Interventions: Drug: Placebo (for L-arginine); Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: L-arginine — 3 gr per day
  Other Names: arginine
  Arms: acetylsalicylic acid and L-arginine
Drug: Placebo (for L-arginine) — 3 gr per day
  Other Names: Magnesia calcined
  Arms: acetylsalicylic acid and placebo
Drug: acetylsalicylic acid — 3 gr per day
  Other Names: aspirin

SUMMARY:
Worldwide, the incidence of preeclampsia ranges from 2 to 10% of pregnancies. The World Health Organization (WHO) estimates that the incidence of preeclampsia is seven times higher in developing countries than in developed (2.8% and 0.4%). In Mexico it is estimated that preeclampsia - eclampsia is a major cause of maternal and perinatal morbidity and mortality. Because it is an idiopathic heterogeneous syndrome associated with endothelial damage, so far there is no effective treatment to decrease the morbidity and mortality of this entity, so it is necessary to strengthen prevention; the use of aspirin alone is inconclusive, in addition to the information the investigators have reduced the effect of these strategies on arterial stiffness; Moreover, it has been observed that L-arginine lowers blood pressure in this population. It is for this that is of interest to know the efficacy and safety of the combination of L-arginine low dose, which is known as an important eNOS in NO production substrate, and aspirin for its qualities of antiinflammatory and anticoagulant in the prevention of preeclampsia and also determine their effect on arterial stiffness as a noninvasive method, as is the applanation tonometry.

DETAILED DESCRIPTION:
It will conduct a clinical trial, double-blind, randomized and placebo control group female patients with 12 weeks of gestation have one or more risk factors for developing preeclampsia. 2 groups will be formed with 82 patients each, chance will determine the intervention (acetylsalicylic + L-arginine acetylsalicylic acid or acid + placebo). At the beginning and end of the intervention clinical and laboratory determinations, the end will be determined in both groups the incidence of preeclampsia, severity and number needed to treat is made. The data obtained were analyzed using SPSS statistical software version 22. It was considered statistically significant at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant before 12 weeks of gestation
* High risk of preeclampsia
* Signature of informed consent in writing

Exclusion Criteria:

* Noncompliance > 20% of drug intake
* Lack of tolerability L-arginine or acetylsalicylic acid
* Compliance with at least one non-inclusion criteria during the course of the study
* Serious adverse event
* Withdrawal of consent

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of preeclampsia | from 20 weeks gestation until 37 weeks
severity of preeclampsia | from 20 weeks gestation until 37 weeks

SECONDARY OUTCOMES:
Pulmonary edema maternal | at week 37
Acute myocardial infarction maternal | at week 37
Stroke maternal | at week 37
Acute respiratory distress syndrome maternal | at week 37
Coagulopathy maternal | at week 37
Renal failure maternal | at week 37
Retinal damage maternal | at week 37
maternal mortality | at week 37
Birth weight | birth
Intrauterine growth restriction | birth
Fetal mortality | birth
systolic blood pressure maternal | from 12 weeks gestation until 37 weeks
diastolic blood pressure maternal | from 12 weeks gestation until 37 weeks
Mean blood pressure maternal | from 12 weeks gestation until 37 weeks
Pulse wave velocity maternal | from 12 weeks gestation until 37 weeks
Adverse effects maternal | from 12 weeks gestation until 37 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leonel García Benavides, PhD, Principal Investigator — University Guadalajara
Locations (1):
- Antiguo Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No